CLINICAL TRIAL: NCT05205057
Title: Salivary Calcium in Post-menopausal Women and Prevalence of Dental Caries
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Other Study IDs: ABSM/EC22/2018
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Salivary Calcium
Keywords: pre-menopausal; Post-menopausal; salivary calcium; dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-menopausal: Pre-menopausal women
  Interventions: Other: Saliva
- Post-menopausal women: post-menopausal women
  Interventions: Other: Saliva

INTERVENTIONS:
Other: Saliva — Unstimulated whole saliva is collected

SUMMARY:
Different phases of a woman's life are puberty, menses, pregnancy, and menopause. Menopause is one of the normal developmental stages in a woman's life, marks the permanent cessation of menstruation. It occurs due to irreversible changes in the hormones.The gradual variation and circulating sex hormones affect women's psychological balance and quality of life. The hormonal changes affect the reproductory system and affect the bone integrity and overall health of the individual. The only source of oocytes in women is an ovary. That is the primary source of oestrogens and progesterone, majorly the androgens. Therefore, various systemic health concerns like vasomotor symptoms, cardiovascular diseases, cancer, sexual problems, osteoporosis, and poor oral health

DETAILED DESCRIPTION:
The presence of estrogen receptors detected through immunohistochemistry in the oral cavity plays a significant role in associating the effect of post-menopausal conditions to variations in the oral environment like salivary hypofunction, oral discomfort, and oral mucosal disorders. The vaginal mucosa and oral mucosa are similar histologically due to stratified squamous epithelium and desquamative growth pattern. Therefore, the variation in hormonal status in post-menopausal women may lead to the proliferation and maturation of oral epithelium in response to circulating estrogens. The keratinocytes and fibroblasts in the gingival tissues are majorly targeted by estrogen leading to periodontitis, fibroblastic hyperplasia, and desquamatic lesions. Therefore, it is a proven fact that gingiva is a traditional estrogen target, leading to the destruction of supporting structures of a tooth, causing periodontitis and thereby exposing tooth structure. Another primary oral manifestation in menopausal women is xerostomia/dryness of the mouth. The salivary components provide defense by maintaining the desired pH and decreasing the prevalence of caries, but estrogen levels directly decrease the salivary flow rate. Thus, the prevalent acidic pH causes demineralization and destruction of enamel, dentin making it more susceptible to dental caries.

A correlation between bone mineral density, salivary calcium levels, and estrogen levels is already established. Hence, the salivary calcium levels can indicate increased demineralization of tooth surface and osteoporosis in menopausal. Hence, the present focuses on estimating salivary calcium levels and their association with the prevalence of dental caries in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* No metabolic disorders
* No medications taken in the past 3 months
* No periodontal disease

Exclusion Criteria:

* Periodontal disease present
* Metabolic disease present
* Medications taken in the past 3 months

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study was conducted among 40 post-menopausal women and 40 premenopausal women reporting to the OPD department of conservative dentistry and endodontics for a regular dental checkup. Individuals with metabolic disorders were and under supplementation were excluded. Women under the age group of 50 - 70 Y were included. Informed consent was obtained, DMFT index was recorded, and unstimulated salivary samples were collected with tarson's collection tubes. Individuals in the case group were further divided into three groups based on their caries experience into group 1: DMFT (D=1); group 2: DMFT(D=2-10), group 3: DMFT <10). The control group included individuals with no caries experience (D=0) and individuals who have not attained their menopause
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Salivary calcium | 2 months
  Salivary calcium change

SECONDARY OUTCOMES:
Dental caries | 2 months
  Dental caries change

CONTACTS AND LOCATIONS:
Locations (1):
- AB shetty Institute of dental sciences, Mangaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
All the results will be shared and attached in the repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years